CLINICAL TRIAL: NCT01645969
Title: A Follow-up Study to Evaluate the One-year Post Treatment Effects of Peginterferon Alfa-2a (PEGASYS) in Patients With HBeAg Positive Chronic Hepatitis B From the Original Study ML 22265
Brief Title: A Follow-Up Study of Patients With HBeAg Positive Chronic Hepatitis B Treated With Pegasys (Peginterferon Alfa-2a) in Study ML22265
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25647
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, prospective, observational study will evaluate the one-year outcomes in HBeAg positive chronic hepatitis B patients who had received Pegasys (peginterferon alfa-2a) in Arm A of study ML22265. Data will be collected from each patient for up to one year post-therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were randomized to study Arm A of ML22265 and were treated and completed follow-up in the study, regardless of treatment response at any time point

Exclusion Criteria:

* Patients unwilling to provide informed consent or abide by the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received treatment and completed follow-up in study arm "A" of study ML22265
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Duration of response (HBeAg seroconversion/HBV DNA reduction/HBsAg loss/seroconversion) after end of treatment | 1 year

SECONDARY OUTCOMES:
Correlation of duration of response with on-treatment response (HBeAg/HBV DNA/HBsAg/ALT) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- China (5):
  - Changsha
  - Fuzhou
  - Guangzhou
  - Wuhan
  - Xi'an